CLINICAL TRIAL: NCT01785394
Title: Changes in Exhaled Breath Temperature During the Pollen Season in Subjects With Allergic Rhinoconjunctivitis Sensitized to Grasses and Effect of Sublingual Immunotherapy
Brief Title: POLlinosis and Exhaled Breath Temperature
Acronym: POLET
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Prof. Todor Popov (Other)
Responsible Party: Sponsor-Investigator, Prof. Todor Popov, Associate Professor, Association Asthma, Bulgaria
Organization: Association Asthma, Bulgaria (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: POLET-12-13
Record Dates: First submitted 2013-02-01; First posted 2013-02-07 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Pollinosis
Keywords: pollinosis; sublingual immunotherapy; exhaled breath temperature
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5 grass allergen extract (Active Comparator): 30 patients will receive the active component 5 grass allergen extract daily during the active pollen season (February-July)
  Interventions: Drug: 5 grass allergen extract
- Placebo (Placebo Comparator): 30 patients will receive placebo
  Interventions: Drug: 5 grass allergen extract

INTERVENTIONS:
Drug: 5 grass allergen extract — 30 patients will be subjected to sublingual immunotherapy with 5 grass allergen extract Staloral, starting with 1 spurt of 10 IR/ml increasing them daily stepwise to 10 spurts, switching then to 1 spurt of 300 IR/ml, increasing daily stepwise to 10 spurts, and then maintaining this dose from February till July. 30 patients will be on placebo.
  Other Names: Staloral

SUMMARY:
The purpose of this study is to determine whether exhaled breath temperature, a surrogate marker of airway inflammation, rises during the pollen season in sensitized subjects with allergic rhinoconjucnctivitis with or without mild asthma. Sublingual Immunotherapy with respective allergens suppresses the seasonal increase of EBT. During the second year (2013) of the trial all patients will be treated with 5 grass allergen extract: carry over differences between the active and placebo arms from the previous year (2012) will be looked for.

DETAILED DESCRIPTION:
Patients with grass pollen allergy are most typical and best responding to sublingual immunotherapy. Their selection will be done in accordance with the criteria listed in Chapter 9 of the World Allergy Organization Position Paper on specific immunotherapy 2009 and in compliance with the rules for good clinical practice.

Proposed primary variable: the difference between the changes of exhaled breath temperature before and in the pollen season of subjects treated with grass-pollen sublingual immunotherapy and the untreated control patients.

Suggested secondary variables: changes over time of exhaled breath temperature in the two groups, difference in symptoms scores, methacholine responsiveness, rescue medication usage.

Statistical analysis: On the basis of the available data about the variability of exhaled breath changes and its changes upon flare up of airway inflammation or after anti-inflammatory treatment we have calculated a sample size of 20 subjects in each group to be sufficient to prove differences in the primary variable with a significance level <0.05. However, as this is "first time ever" type of pilot study on sublingual immunotherapy and exhaled breath temperature in grass-pollen patients, this estimate is relative. By all means this study will identify trends to be used for sample size calculations in future studies. During the second year of the study when all patients will be on active treatment with 5 grass allergen extract, carry over effects from the first year of treatment with 5 grass allergen extract or placebo on exhaled breath temperature will be explored.

ELIGIBILITY:
Inclusion Criteria:

* 60 randomized patients from either sex
* age range 5-55 years
* included patients should have a proven grass pollen sensitization

Exclusion Criteria:

* age under or above the stated
* lack of any other concomitant allergen sensitivities that may blur the clinical course of the natural exacerbation due to pollen

Ages: 5 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Changes of exhaled breath temperature before and during the pollen season of subjects treated with 5 grass allergen extract sublingually and the untreated control patients. | 6 months in year 1 (2012): baseline and at month 6; and 6 months in year 2 (2013): baseline and month 6.
  The primary objective of the study is to evaluate the differences between the changes of exhaled breath temperature before and in the pollen season of subjects treated with 5 grass allergen extract applied sublingually and untreated control patients. Possible carry-over differences between the same two arms will be explored during the second year of the trial. Calculations will involve difference between assessment at month 6 and baseline for year 1 (2012) and in year 2 (2013) and comparisons between the two arms of the study will be made.

SECONDARY OUTCOMES:
Effect of the treatment on symptoms and objective measurements in blood | 6 months in year 1 (2012): baseline and at month 6; and 6 months in year 2 (2013): baseline and month 6.
  Changes over time of exhaled breath temperature in the two groups, difference in symptoms scores, methacholine responsiveness, rescue medication usage, changes in blood cell counts, C-reactive protein, IL13 and periostin will be calculated (difference between assessment at month 6 and baseline) for year 1 (2012) and Year 2 (2013) and compared between the two arms of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Todor Popov, MD, PhD, Principal Investigator — Professor of Allergology
Locations (1):
- Medical University Sofia, Department of Allergology, Sofia, Bulgaria

REFERENCES:
- [Background] Xepapadaki P, Xatziioannou A, Chatzicharalambous M, Makrinioti H, Papadopoulos NG. Exhaled breath temperature increases during mild exacerbations in children with virus-induced asthma. Int Arch Allergy Immunol. 2010;153(1):70-4. doi: 10.1159/000301581. Epub 2010 Apr 1. PMID 20357487
- [Background] Popov TA, Kralimarkova T, Tzachev C, Dimitrov V, Mun KK, Gill J. Exhaled breath temperature measurement made easy. Pediatr Allergy Immunol. 2009 Mar;20(2):200-1; author reply 202-3. doi: 10.1111/j.1399-3038.2008.00837.x. Epub 2008 Nov 10. No abstract available. PMID 19017281
- [Background] Popov TA, Dunev S, Kralimarkova TZ, Kraeva S, DuBuske LM. Evaluation of a simple, potentially individual device for exhaled breath temperature measurement. Respir Med. 2007 Oct;101(10):2044-50. doi: 10.1016/j.rmed.2007.06.005. Epub 2007 Jul 12. PMID 17624752
- [Background] Braunstahl GJ, Hellings PW. Nasobronchial interaction mechanisms in allergic airways disease. Curr Opin Otolaryngol Head Neck Surg. 2006 Jun;14(3):176-82. doi: 10.1097/01.moo.0000193186.15440.39. PMID 16728896
- [Derived] Kralimarkova TZ, Popov TA, Staevska M, Mincheva R, Lazarova C, Racheva R, Mustakov TB, Filipova V, Koleva M, Bacheva K, Dimitrov VD. Objective approach for fending off the sublingual immunotherapy placebo effect in subjects with pollenosis: double-blinded, placebo-controlled trial. Ann Allergy Asthma Immunol. 2014 Jul;113(1):108-13. doi: 10.1016/j.anai.2014.03.019. Epub 2014 Apr 16. PMID 24745701